CLINICAL TRIAL: NCT02943408
Title: Development of a Patient Centered Mental Health Intervention for Recent Veterans
Acronym: PCC MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2159-W; 1IK2RX002159-01A2 (NIH)
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Anxiety; Substance-Related Disorders
Keywords: Veterans; mental health; Patient-Centered Care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Substance-Related Disorders; Psychological Well-Being | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to participant intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- person-centered mental health intervention (PCMHI) (Experimental): We anticipate that the PCMHI will be comprised of three, one-hour sessions offered over three to six weeks, scheduled at the participants' preference. Sessions will be one-on-one and the peer support specialist interventionist.
  Interventions: Behavioral: person-centered mental health intervention
- health and wellness (Active Comparator): The control condition will be an educational health and wellness intervention for stress related disorders that will match the experimental condition for time and attention. The control condition will be three, one hour, individual sessions covering the symptom cycle, managing stress, and identifying social supports.
  Interventions: Behavioral: health and wellness

INTERVENTIONS:
Behavioral: person-centered mental health intervention — We anticipate that the PCMHI will be comprised of three, one-hour sessions offered over three to six weeks, scheduled at the participants' preference. Sessions will be one-on-one and the peer support specialist interventionist.
  Arms: person-centered mental health intervention (PCMHI)
Behavioral: health and wellness — The control condition will be an educational health and wellness intervention for stress related disorders that will match the experimental condition for time and attention. The control condition will be three, one hour, individual sessions covering the symptom cycle, managing stress, and identifying social supports.
  Arms: health and wellness

SUMMARY:
Recent Veterans of the OIF/OEF/OND conflicts are presenting in VA care with high rates of: PTSD, depression, anxiety, and alcohol abuse, reporting significant difficulties with community reintegration, and dropping out of mental health care at high rates. Surveys of recent Veterans show that Veterans want the VA to provide mental health care tailored to their concerns and reintegration priorities. The VA is committed to providing personalized, proactive, patient centered care (PCC); but little research or intervention development has been done on PCC in mental health care settings and preliminary research indicates Veterans may lack the skills and knowledge to be active partners in PCC. This study aims to examine PCC behaviors in VA mental health care and, informed by this data, develop a brief patient centered mental health intervention that will help recent Veterans take the lead in their care personalization and support their functional recovery. Results from this study will demonstrate the acceptability, feasibility, and preliminary efficacy of this intervention.

DETAILED DESCRIPTION:
Project Background: The term "recent Veterans" refers to Veterans who served in the military operations Operation Enduring Freedom, Operation Iraqi Freedom, and Operation New Dawn. Almost 60% of recent Veterans who received VA care have been diagnosed with a mental health disorder, most commonly posttraumatic stress disorder (32%), depressive disorders (26%), anxiety disorders (25%), and substance abuse (13%). The research literature consistently confirms that recent Veterans with stress-related mental health disorders experience impairment in functional domains of health (overcoming and managing disease), purpose (meaningful daily activities and participation in society), and community (positive relationships and social networks).

Project Objectives: The proposed research will characterize patient centered care in VA mental health care and produce a brief patient centered intervention that will empower Veterans to lead and personalize their mental health care in support of their functional recovery. In Aim 1 of this research the investigators will characterize rates of providers' and recent Veterans' (n=30) participation in the four components of PCC, as well as barriers and facilitators of each PCC component, to inform development of a brief patient centered mental health intervention in Aim 2. In Aim 2 the investigators will develop a brief patient centered mental health intervention for recent Veterans experiencing stress-related mental health disorders and conduct a pre-pilot demonstration (n=10) to assess acceptability. This intervention will be informed by data collected in Aim 1 and developed using an iterative process of discussion with and input from recent Veterans, VA mental health providers, peer specialists, and researchers. Finally in Aim 3 the investigators will test the feasibility and preliminary efficacy of the brief intervention by conducting a randomized controlled trial with 48 recent Veterans with stress-related mental health disorders.

Project Methods: In Aim 1 data will be collected at one time point using surveys and a recording of a Veteran provider encounter which will be coded to quantify Veteran and provider patient centered care behaviors. Intervention development in Aim 2 will be led by a multi-stakeholder Advisory Panel and further developed using Veteran focus groups. Acceptability will be demonstrated via qualitative interviews following a pre-pilot demonstration project with 10 Veteran participants. In Aim 3 data will be collected at baseline, post-RCT participation, and 3 month and 6 month follow-up. Feasibility will be assessed with study administration data on engagement and participation in the intervention and preliminary efficacy will be evaluated via quantitative analysis of functioning from self-report surveys.

Note: Measure of Patient Centered Care (Patient-centered Communication) was removed as a measure. The MPCC requires recording a patient-provider encounter and coding it. When the pandemic occurred previous methods of recording encounters and physically bringing an approved recording device to the provider's office prior to the session, was no longer viable. Investigators had to suspend recording until approved technology guidance was provided. When a means was identified it was so cumbersome no providers agreed to record.

ELIGIBILITY:
Inclusion Criteria:

Per medical record review:

* military service in Operation Iraqi Freedom, Operation Enduring Freedom, or Operation New Dawn (OIF/OEF/OND)
* Veteran accessed mental health care (MHC) service at designated study site for the first time in the last 6 months OR the first time in the last 6 months after at least a one year gap in mental health care
* have a diagnosis of PTSD (309.81), major depressive disorder (296.20-296.23, 296.30-296.33), other specified or unspecified depressive disorder (311), social anxiety disorder (300.23), panic disorder (300.01), generalized anxiety disorder (300.02), other specified or unspecified anxiety disorder (300.09, 300.00), substance use disorders (303.90, 304.00, 304.10, 304.30), Unspecified Trauma and Stressor-Related Disorder (309.9), Other Specified Trauma and Stressor-Related Disorder (309.89), or Adjustment Disorder (309.20- 309.25)
* age between 18 and 65
* sufficient clinical stability to participate as deemed by a treatment provider
* Veteran consents to having one mental health encounter recorded and coded
* Veteran's relevant provider consents to having one mental health encounter recorded and coded

Exclusion Criteria:

Per medical record review:

* current diagnosis of a psychotic disorder meeting criteria established by the VA Serious Mental Illness Treatment, Research, and Evaluation Center (SMITREC):

  * schizophrenic disorders (295.0-295.9)
  * affective psychoses (296.0-296.1, 296.4-296.8)
  * or major depression with psychotic features (296.24, 296.34)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hack, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (3):
- United States (3):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - Perry Point VA Medical Center VA Maryland Health Care System, Perry Point, MD, Perry Point, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Final datasets will be maintained locally until enterprise-level resources become available. Final data sets will be made available to the public upon request as outlined in Question 5 above. Specifically, complete person-level data will be provided as either a Limited Dataset or as a de-identified, anonymized dataset depending on the needs of the requester.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Started | 24 | 24
Baseline | 24 | 23
Time Point 2 : 4-7 Weeks Post Baseline | 21 | 19
Time Point 3: 3 Months Post Time Point 2 | 21 | 22
Completed | 17 | 22
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (8.1) | 40.5 (9.1) | 39.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 11 | 4 | 15
  White | 10 | 16 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 47
Veterans RAND 36-Item Health Survey - role limitations due to emotional problems [Mean (Standard Deviation); unit: score on a scale] — Scores range from 0 to 100 with higher scores indicating better functioning
  score on a scale | 47.57 (26.18) | 47.10 (23.52) | 47.34 (26.64)
Veterans RAND 36-Item Health Survey - vitality [Mean (Standard Deviation); unit: score on a scale] — Scores range from 0 to 100 with higher scores indicating better functioning
  score on a scale | 25.42 (21.51) | 27.83 (18.88) | 26.60 (20.08)
Veterans RAND 36-Item Health Survey - social functioning) [Mean (Standard Deviation); unit: score on a scale] — Scores range from 0 to 100 with higher scores indicating better functioning
  score on a scale | 35.42 (29.64) | 29.35 (20.51) | 32.45 (25.49)
Veterans RAND 36-Item Health Survey - mental health [Mean (Standard Deviation); unit: score on a scale] — Scores range from 0 to 100 with higher scores indicating better functioning
  score on a scale | 40.83 (22.10) | 46.61 (20.95) | 43.66 (21.51)
World Health Organization Disability Assessment Schedule 2.0 - household life activities [Mean (Standard Deviation); unit: score on a scale] — Items are scored on a 0-100 scale. Lower scores indicate less disability
  score on a scale | 57.92 (25.70) | 59.57 (26.02) | 58.72 (25.59)
World Health Organization Disability Assessment Schedule 2.0 - school/work life activities [Mean (Standard Deviation); unit: score on a scale] — Items are scored on a 0-100 scale. Lower scores indicate less disability
  score on a scale | 46.83 (28.70) | 42.86 (19.69) | 44.96 (24.59)
World Health Organization Disability Assessment Schedule 2.0 - participation in community activities [Mean (Standard Deviation); unit: score on a scale] — Items are scored on a 0-100 scale. Lower scores indicate less disability
  score on a scale | 56.60 (23.02) | 57.34 (21.67) | 56.94 (22.28)

OUTCOME MEASURES:

1. Primary Outcome: Veterans RAND 36-Item Health Survey (Change in Self-assessment of Functioning - Role Limitations) Due to Emotional Problems
Description: The Veterans RAND 36-Item Health Survey measures health-related quality of life in 8 domains, 4 of which will be utilized in this study: (1) role limitations due to emotional problems, (2) vitality, (3) social functioning, and (4) mental health. Scores range from 0 to 100 with higher scores indicating better functioning.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 50.98 (29.3) | 47.35 (27.38)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .90, Mixed Models Analysis

2. Primary Outcome: Veterans RAND 36-Item Health Survey (Change in Self-assessment of Functioning - Vitality)
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 29.12 (24.25) | 28.64 (17.61)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .99, Mixed Models Analysis

3. Primary Outcome: Veterans RAND 36-Item Health Survey (Change in Self-assessment of Functioning - Social Functioning)
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 46.32 (33.88) | 36.36 (25.27)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .56, Mixed Models Analysis

4. Primary Outcome: Veterans RAND 36-Item Health Survey (Change in Self-assessment of Functioning - Mental Health)
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 50.82 (23.65) | 48.55 (24.33)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .85, Mixed Models Analysis

5. Primary Outcome: World Health Organization Disability Assessment Schedule 2.0 (Change in Self-assessment of Functioning - Household Life Activities)
Description: World Health Organization Disability Assessment Schedule 2.0 is a 36-item assessment of health and disability across physical and mental health disorders in both clinical and non-clinical settings/populations. It closely corresponds with the International Classification of Functioning, Disability, and Health (ICF). Subscales measuring (1) life activities such as domestic responsibilities, (2) life activities such as school and work, and (3) participation in community activities. Items are scored on a 0-100 scale. Lower scores indicate less disability.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 41.18 (24.47) | 50 (23.71)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .43, Mixed Models Analysis

6. Primary Outcome: World Health Organization Disability Assessment Schedule 2.0 (Changes in Self-assessment of Functioning - School/Work Life Activities)
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 36.26 (30.23) | 39.52 (23.98)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .82, Mixed Models Analysis

7. Primary Outcome: World Health Organization Disability Assessment Schedule 2.0 (Changes in Self-assessment of Functioning - Participation in Community Activities)
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 41.91 (24.32) | 48.86 (21.79)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .50, Mixed Models Analysis

8. Secondary Outcome: Depression Anxiety Stress Scale-21 (Change in Depression Symptoms)
Description: Depression Anxiety Stress Scale is 21 self report items scored on a 4-point Likert scale that ranges from 0 (not at all) to 3 (applied very much). It has three subscales: depression (7 items with a possible score from 0 to 21), anxiety (7 items with a possible score from 0 to 21), and stress (7 items with a possible score from 0 to 21). Higher scores indicate greater symptomology.
Time Frame: 6 months
Population: participants who completed a DASS-21 at 6 months post baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 7.77 (5.72) | 8.55 (6.05)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .56, Mixed Models Analysis

9. Secondary Outcome: Depression Anxiety Stress Scale-21 (Change in Anxiety Symptoms)
Description: as for outcome 8
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 6.77 (5.15) | 8.23 (5.96)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .92, Mixed Models Analysis

10. Secondary Outcome: PTSD Checklist for DSM-5 (Change in PTSD Symptoms)
Description: PTSD Checklist for DSM-5 is the most current version of the PTSD Check List (PCL), the gold standard of PTSD symptom assessments. Its 20-items use a 5-point Likert scale (0-not at all to 4-extremely) that maps on to the diagnostic criteria outlined in the DSM-5. The PCL-5 is appropriate for both clinical and research purposes and is recommended for monitoring symptom change. The PCL-5 is summed to create a total score with a possible range of 0 to 80. A score of 31-33 or higher is indicative of a provisional diagnosis of PTSD and preliminary validation has established that a 10 point change is clinically significant.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 31.65 (16.19) | 38.55 (21.59)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .65, Mixed Models Analysis

11. Secondary Outcome: Alcohol Use Disorders Identification Test (Change in Alcohol Use Symptoms)
Description: Alcohol Use Disorders Identification Test is a 10-item self-report instrument with each item scored on a scale of 0-4 for a total possible score of 0 to 40. The items obtain information on the frequency and amount of drinking and alcohol-related problems. A score of 8 or more is associated with harmful or hazardous drinking.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 17 | 22
score on a scale | 3 (4.12) | 4.36 (4.01)
Statistical Analysis 1: Comparison: Person-centered Mental Health Intervention (PCMHI) vs Health and Wellness; Test type: Superiority; p = .35, Mixed Models Analysis

12. Secondary Outcome: Drug Abuse Screening Test (DAST-10) - (Change in Substance Use Symptoms)
Description: Drug Abuse Screening Test (DAST) is a 10 item, yes or no response measure of drug use. The possible scores range from 0 to 10. The DAST 10 scores are divided into five levels of symptomology (0 No problems reported; 1-2 Low; 3-5 Moderate; 6-8 Substantial; 9-10 Severe) and level change is considered clinically significant.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
Number analyzed (Participants) | 24 | 24
units on a scale | .63 (1.56) | .74 (1.29)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Person-centered Mental Health Intervention (PCMHI) | Health and Wellness
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
* This was a pilot randomized controlled trial so the sample size is small.
* Approximately one third of the way through recruitment and randomization the COVID-19 pandemic began. This caused disruption to the data collection process and required the interventions to transition from in-person to telehealth platforms. We were not able to record patient-provider encounters to code with the Measure of Patient Centered Communication. Therefore, no results for that measure are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02943408/Prot_SAP_000.pdf